CLINICAL TRIAL: NCT03830723
Title: Effect of Personalized Dosages of Rekovelle on the Number of Mature Follicles Reached in Intra-uterine Insemination
Brief Title: Personalized Insemination Treatment Study
Acronym: PITS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ovord
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-01

CONDITIONS: Infertility; Intrauterine Insemination; Reproduction
MeSH Terms: conditions — Infertility | interventions — follitropin delta

STUDY DESIGN:
Intervention Model Description: open-label, prospective, dose-finding, single centre pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rekovelle (Follitropin delta) (Other): All participants will receive a prescription for study medication Rekovelle (follitropin delta)
  Interventions: Drug: Follitropin delta

INTERVENTIONS:
Drug: Follitropin delta — Study medication doses during all 3 insemination will be personalized using a suggested algorithm
  Other Names: Rekovelle

SUMMARY:
This study is intended for women undergoing their first cycle of 3 intrauterine inseminations. All 3 inseminations will be personalized by using algorithms to determine the dose of study medication.

DETAILED DESCRIPTION:
Study medication dosage for the first insemination cycle will be based on the woman's age as well as her Anti-Mullerian Hormone (AMH) levels.

Study medication dosage for the second and third insemination will depend on ovarian response (number of follicles) during previous insemination cycle and woman's age

ELIGIBILITY:
Inclusion Criteria:

* Women having consented to the study
* Women followed at fertility center
* First IUI cycle
* Women between the ages of 18 to 42 inclusively at time of consent form signature
* AMH < 35 pmol/L (4.9 ng/mL) in participants' file in the last 24 months
* At least one permeable Fallopian tube confirmed by laparoscopy, hysterosalpingography (HSG), hysterosalpingosonography (HSSG) or one pregnancy in the last 3 years
* Insemination with either partner or donor sperm
* Male partner semen analysis considered adequate for IUI in accordance to the centre's standard practice
* Menstrual cycles from 26 to 39 days
* Presence of both ovaries

Exclusion Criteria:

* Unable to consent
* Body weight >100 kg
* AMH ≥35 pmol/L (4.9 ng/mL) in participants' file in the last 24 months
* Severe malformation (unicornuate or bicornuate uterus) or uterine anomaly including fibroids ≥ 5 cm
* Uncontrolled thyroid or adrenal dysfunction
* Pituitary tumour
* Persistent ovarian cysts or enlargement not due to PCOS (Polycystic ovary syndrome) > 3 cm
* Anovulatory women
* Use of contraceptives in the last 3 months prior to start of stimulation
* Diagnosis of hydrosalpinx
* Malignancies
* Breast pathology incompatible with gonadotropin stimulation
* Hypersensitivity to follitropin delta or to any ingredient in the formulation
* Addition of other infertility medication that can influence follicle stimulation and maturation such as growth hormone (GH)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Fertile women undergoing intrauterine insemination
Enrollment: 110 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Ovarian response | 1 year
  Evaluate the dose-response Relationship of Rekovelle with respect to ovarian response in participants undergoing controlled ovarian stimulation for intrauterine insemination

SECONDARY OUTCOMES:
Pregnancy rate | 1 year
  Evaluate pregnancy rate 6-8 weeks after insemination by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No